CLINICAL TRIAL: NCT04492280
Title: Evaluation of the Role of Hydrocortisone Either Alone or Combined With Fludrocortisone in the Outcome of Septic Shock in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona Ammar, Assistant Professor of Anesthesia and Intensive Care, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 176/2018
Record Dates: First submitted 2020-07-17; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Hydrocortisone; Fludrocortisone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. Group H (Active Comparator): These patients will receive standard therapy for sepsis plus Hydrocortisone (Solucortef®, E.I.P.I.co. under license of Pfizer) at dose 50mg every 6 hours by Intra venous route.
  Interventions: Drug: Hydrocortisone
- 2. Group HF (Active Comparator): These patients will receive standard therapy for sepsis plus Hydrocortisone (Solucortef®) at dose of 50mg every 6 hours by Intra venous route and Fludrocortisone (Cortilon®, Amoun) 50 Microgram once daily by nasogastric tube for one week
  Interventions: Drug: Hydrocortisone
- 3. Group C (Placebo Comparator): These patients will receive standard therapy for sepsis.
  Interventions: Drug: Hydrocortisone

INTERVENTIONS:
Drug: Hydrocortisone — After approval of the ethical committee of faculty of Medicine Ain Shams University and obtaining a written informed consent from all patients or their legal guardians, the study will be conducted on 66 patients subdivided randomly via computer closed envelopes method into 3 equal groups, 22 patients for each group; group HF (hydrocortisone & fludrocortisone), group H (hydrocortisone) and group C (control group).
  Other Names: Fludrocortisone

SUMMARY:
During Infection, oflfending microbes interact with the host immune system producing a downstream inflammatory cascade involving cytokines and other mediators, which in turn triggers a systemic response. The resultant effects linclude vasodilation, increased vascular permeability, myocardial depression, and impairment of the coagulation cascade, resulting in global imbalance of systemic oxygen supply and demand. During the late stage of sepsis, immunosuppression predominates, leading to multi-organ dysfunction and further clinical deterioration .

Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection with two or three on Quick Sepsis-related organ failure assessment score (qSOFA). Septic shock is defined as the presence of sepsis and refractory hypotension to fluid management. Vasopressors are needed to maintain systolic blood pressure more than 90mmHg or mean blood pressure more than 65 mmHg .

Experimental and Clinical evidence suggests that sepsis is associated with dysregulated response of Hypothalamic-pituitary-adrenal axis that may involve any of the steps from cortisol production to cortisol use by cells .

Glucocorticoid therapy for the treatment of septic shock remains controversial, with conflicting evidence regarding a mortality benefit. It has been used in patients with septic shock who remained hypotensive after fluid and vasopressor resuscitation.

Fludrocortisone is a corticosteroid and acts as a powerful mineralocorticoid along with some additional but comparatively very weak glucocorticoid activity. Relative to cortisol, it is to 10 times the glucocorticoid potency but 250 to 800 times the mineralocorticoid potency .

Fludrocortisone is added to hydrocortisone to provide additional mineralocorticoid potency. The rationale for adding mineralocorticoid treatment is that an experimental sepsis study showed marked nuclear factor NF-κB mediated down regulation of vascular mineralocorticoid receptors .

Corticosteroids attenuate inflammation in various organs an effect partly related to inhibition of nuclear factor NF-κB. Improve cardiovascular function by restoring effective blood volume through increased mineralocorticoid activity and by increasing systemic vascular resistance through vascular α-Adrenergic responsiveness and reduces inflammation-mediated vasodilation .

ELIGIBILITY:
Inclusion Criteria:

* This study will be conducted on patients between 18-80 years old, both sexes who are suffering from septic shock and have any of the following any of 1, 2, or 3 criteria
* CLINICAL EVIDENCE OF INFECTION WITHIN THE PREVIOUS 72 HOURS OF ICU ADMISSION (any of a, b, or c)

  1. Presence of polymorphonuclear cells in a normally sterile body fluid.
  2. Culture or Gram stain of blood, sputum, urine or normally sterile body fluid positive for a pathogenic micro-organism.
  3. Focus of infection identified by visual inspection (e.g. ruptured bowel with the presence of free air or bowel contents in the abdomen found at the time of surgery, wound with purulent drainage).
* Sepsis-related organ failure assessment (SOFA) score of 3 or 4 (on a scale of 0 to 4 for each of six organ systems) for at least 2 organs and at least 6 hours (Singer et al., 2016).
* Vasopressors Therapy ( norepinephrine , epinephrine , or any other vasopressors at a dose of ≥ 0.25 µg / kg / minute ) for at least 6 hours to maintain a systolic blood pressure of at least 90 mm Hg or mean blood pressure of at least 65 mm Hg (Singer et al., 2016).

Exclusion Criteria:

* Refusal of patient or legal guardian to consent to participate in the study.
* Pregnancy and lactation.
* Gastrointestinal Bleeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
• Mortality rate due to septic shock as a cause. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Mona A Ammar, Cairo, Egypt